CLINICAL TRIAL: NCT03617094
Title: Early Percutaneous Vertebroplasty Versus Standard Conservative Treatment in Thoracolumbar Vertebral Fractures. Monocentric, Prospective, Randomised and Compared Clinical Study
Brief Title: Early Percutaneous Vertebroplasty Versus Standard Conservative Treatment in Thoracolumbar Vertebral Fractures
Acronym: AGIL11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 38RC17.276
Record Dates: First submitted 2018-05-28; First posted 2018-08-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Vertebral Fracture
Keywords: Vertebral fracture; Early Percutaneous Vertebroplasty; Standard Conservative Treatment; Kyphosis angle
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early percutaneous vertebroplasty (EPV) (Experimental): Surgical procedure of percutaneous vertebroplasty.
  Interventions: Device: Early percutaneous vertebroplasty (EPV)
- Standard Conservative treatment (CT) (Active Comparator): Thoracolumbar corset.
  Interventions: Device: Standard Conservative treatment (CT)

INTERVENTIONS:
Device: Early percutaneous vertebroplasty (EPV) — Treatment consists of percutaneous acrylic bone cement injection using a trocar under scope control and general anesthesia.
  Arms: Early percutaneous vertebroplasty (EPV)
Device: Standard Conservative treatment (CT) — Treatment consists of using a made-to-measure 3 point thoracolumbar corset,that is worn for 3 months: night and day during the first 6 week period of the treatment, and then only the day for the next 6 week period.
  Arms: Standard Conservative treatment (CT)

SUMMARY:
The aim of this study is to evaluate the efficacy of carrying out early vertebroplasty procedure, compared to the standard conservative treatment (corset), in order to prevent residual deformations that could occur in complications of vertebral fractures that are medically treated using a corset.

This is a monocentric, randomized, parallel group, prospective and open-label study.

DETAILED DESCRIPTION:
In this study, 58 patients with a vertebral fracture no more than 10 days old (with a max of 15 days old) will be enrolled. Treatment will be randomly allocated in 2 groups: Early percutaneous vertebroplasty (EPV group) or standard conservative treatment (corset, CT group). Patients will be followed up during 3 months after treatment. They will receive standard care for a vertebral fracture at the Grenoble-Alpes University Hospital.

Evaluated criteria: Vertebral kyphosis evolution, Pain, Efficacy and Quality of vertebroplasty procedure, Tolerance and observance of the standard treatment, Safety, Physical performance, Quality of life, Autonomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Fracture localisation : vertebrae from T8 to L5
* Recent fracture (< 10 days, maximum 15 days)
* CT scan showing a fracture of the superior endplate and of the anterior cortex of the vertebral body of type A1 according to the Magerl classification AND vertebral kyphosis deformation < 30°
* Patient affiliated to the French social security system or an equivalent system
* Patient who has signed consent form

Exclusion Criteria:

* Multiple level fracture
* Repeated fracture at the same level
* Others peripheral fractures
* Contraindication for percutaneous procedure
* Contraindication for vertebroplasty procedure (pathology with risk of decompensation, coagulation problems, deformation considered by the surgeon to be inaccessible by vertebroplasty procedure, presence of an infected site)
* Contraindication for anasthesia
* Methylmethacrylate (MMA) allergy known
* Impossibility to plan the start of the treatment (set up of treatment or carrying out of a vertebroplasty gesture) within a maximum deadline of 15 days after the fracture
* Body Mass Index (BMI) > 31,5
* Progressive local infection
* Progressive local cancer
* Patient presenting cognitive disorder with behavioural disorder which could disturb the treatment
* Non-cooperative patient
* Patient who can not be followed up at Grenoble hospital during the 3 months of the study
* Patient concerned by articles L1121-5, L1121-6, L1121-8 of the French public health code

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Vertebral kyphosis change between fracture diagnosis and after 3 months of treatment, in the two groups | Diagnosis, and after 3 months of treatment
  Difference in the kyphotic angle measured at the fracture diagnosis and after 3 months of treatment

SECONDARY OUTCOMES:
Compare the pain evolution between fracture diagnosis and after 3 months of treatment, in the two groups | diagnosis, after 24 hours, 45 days and 3 months of treatment
  Pain will be assessed using a Visual Analogic Scale (score from 0 to 10)
Evaluation of the efficacy of early vertebroplasty procedure (EPV arm) - Kyphotic Angle | Diagnosis, immediat post-op, after 45 days and 3 months of treatment
  Kyphotic angle (KA)
Evaluation of the efficacy of early vertebroplasty procedure (EPV arm) - Anterior vertebral height | Diagnosis, immediat post-op, after 45 days and 3 months of treatment
  Anterior vertebral height (HA)
Evaluation of the efficacy of early vertebroplasty procedure (EPV arm) - Vertebral Compression Ratio | Diagnosis, immediat post-op, after 45 days and 3 months of treatment
  Vertebral Compression Ratio (AP)
Evaluation of the efficacy of early vertebroplasty procedure (EPV arm) - Regional kyphotic angle | Diagnosis, immediat post-op, after 45 days and 3 months of treatment
  Regional kyphotic angle (RA)
Quality of the early vertebroplasty procedure (EPV arm) assessed as the quality of cement filling | Immediately post-op
  Evaluation of the quality of cement filling as poor / acceptable / satisfactory, according to the method described in L.Garnier and col, 2012.
Tolerability of the treatment by corset (CT arm) assessed using the number of thoracolumbar corset readjustments during treatment | 3 months
  Number of thoracolumbar corset readjustments carried out during follow up (3 months)
Evaluation of the observance of the treatment by corset (CT arm) | 3 months
  Daily observance report of thoracolumbar corset wear during follow up (3 months)
Comparison of the adverse events during the study between the two groups | 3 months
  Numbers of adverse events (classification : minor, mild, severe)
Comparison of physical performance evolution between 24h and 3 months after treatment, between the two groups | 24 hours and 3 months after treatment
  Physical performance will be assessed using Short Physical Performance Battery test (SPPB, score from 0 to 12)
Comparison of the evolution in the autonomy of the patients using ADL questionnaire (before and after vertebral fracture, and 3 months after treatment), between the two groups | Diagnosis (before / after fracture), and 3 months after treatment
  ADL (Activities of Daily living) questionnaire score
Comparison of the evolution in the autonomy of the patients using IADL questionnaire (before and after vertebral fracture, and 3 months after treatment), between the two groups | Diagnosis (before / after fracture), and 3 months after treatment
  IADL (Instrumental ADL) questionnaire score
Comparison of the evolution of quality of life using SF-36 questionnaire score (before and after vertebral fracture, and 3 months after treatment) between the two groups | Diagnosis (before / after fracture), and 3 months after treatment
  SF-36 (Short Form-36 Health Survey) questionnaire score
Comparison of the evolution of quality of life using QUALEFFO questionnaire (before and after vertebral fracture, and 3 months after treatment) between the two groups | Diagnosis (before / after fracture), and 3 months after treatment
  QUALEFFO (Quality of life questionnaire of the European Foundation for Osteoporosis) questionnaire score
Comparison of the number of days of hospitalization between the two groups | 3 months
  Length of hospitalization (days)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Boudissa, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, Grenoble, France

REFERENCES:
- [Background] Garnier L, Tonetti J, Bodin A, Vouaillat H, Merloz P, Assaker R, Court C; French Society for Spine Surgery. Kyphoplasty versus vertebroplasty in osteoporotic thoracolumbar spine fractures. Short-term retrospective review of a multicentre cohort of 127 consecutive patients. Orthop Traumatol Surg Res. 2012 Oct;98(6 Suppl):S112-9. doi: 10.1016/j.otsr.2012.03.018. Epub 2012 Aug 28. PMID 22939104